# COVER PAGE

HOPE Intervention for COVID-19 NCT04376515 6/8/2021

# University of California, Irvine Study Information Sheet

## Harnessing Online Peer Education (HOPE) COVID-19 Vaccine Study

## **Lead Researcher**

Sean Young, PhD
Department of Emergency Medicine, Department of Informatics
714-456-5239
syoung5@uci.edu

- Please read the information below and ask questions about anything that you do not understand. A researcher listed above will be available to answer your questions.
- You are being asked to participate in a research study. Participation in this study is voluntary. You
  may choose to skip a study procedure, refuse to participate, or discontinue your involvement at any
  time without penalty or loss of benefits. You are free to withdraw from this study at any time. If you
  decide to withdraw from this study you should notify the research team immediately.
- You are being asked to participate in this research study to study whether peer leaders in an online social network can help to teach participants about risks, prevention methods, and promote the use of vaccines to help stop the spread of COVID-19.
- You are eligible to participate in this study if you meet the following inclusion criteria:

#### Inclusion criteria:

- 1. Adults, 18+, who are competent to give informed consent
- 2. English speakers only
- 3. U.S. Resident
- 4. Part of phase 1a or 1b of COVID-19 vaccine rollout healthcare personnel and frontline essential workers (employment verified through LinkedIn profile or similar)
- 5. Uses social media and/or online communities greater than twice per week
- 6. Has, or is willing to accept a friend request and group invite from our Facebook social media page
- 7. Has not received a COVID-19 vaccine and does not have medical conditions or other circumstances preventing them from receiving one
- **Phase 1a** includes **healthcare personnel** such as physicians, nurses, technicians, therapists, pharmacists, administrative staff, environmental services staff, students, and other trainees.
- Phase 1b includes frontline essential workers such as fire fighters, police officers, corrections
  officers, food and agricultural workers, United States Postal Service workers, manufacturing workers,
  grocery store workers, public transit workers, and those who work in the educational sector
  (teachers, support staff, and daycare workers.)
- See CDC recommendations for further details: <a href="https://www.cdc.gov/coronavirus/2019-ncov/vaccines/recommendations.html">https://www.cdc.gov/coronavirus/2019-ncov/vaccines/recommendations.html</a>
- The research procedures involve the following:
  - 1. Fill out an online questionnaire (baseline and at 4-weeks; approximately 15 minutes each) assessing your knowledge, attitudes, and behaviors in regards to COVID-19/COVID-19 virus. You will also have the option to email us to receive resources about COVID-19 vaccination.

- 2. If on any surveys, you respond that you have received the vaccine, we will invite you text/email us a picture of your vaccine card.
- 3. Join the HOPE UCI Facebook/social media page and group. You will be assigned to an online group. Participants (and peer leaders if you are in the intervention group) may request to become your Facebook "friends" and to chat with you. You may be invited to follow us on other social media like TikTok. Other participants (and peer leaders if you are in the intervention group) may request to follow you on other social media and interact with you. If your settings allow, we will track your social networks to see how they change and grow.
- 4. You will be asked to log onto the Facebook group page at least 3 times a week for 4 weeks. However, this participation is voluntary.
- 5. Each week of the 4-week intervention, we might take screenshots of your social networks to measure social network metrics like number of shared friends and distance between friends. We might also ask you to allow us to access your social network data by allowing access to an analytic application (e.g. Facebook Connect application, TikTok Pro Account) or other software used by social network researchers that connects to online social networks and allows you to grant access to researchers recording social network dynamics.
- Possible risks/discomforts associated with the study include the following:
  - Risks of breach of confidentiality. While the research team will do their best to maintain confidentiality, including coding any identifiable data, and storing data on an secure server, the nature of a Facebook group is such that we cannot guarantee complete confidentiality due to the possibility, although it may be discouraged, of group members disclosing information discussed in the group.
  - Emotional risk. Coronavirus is currently a sensitive topic and has caused many people anxiousness and stress. Talking about this topic may trigger an unwanted emotional response.
- Participating in this study may help you gain an understanding of healthy behaviors. The results of the research may also benefit society by educating others about health and promoting COVID-19 vaccination.
- There are no alternative procedures available. The only alternative is not to participate in this study.
- Your participation will be compensated in the form of an online Amazon gift certificate. Provided you are eligible after verifying your LinkedIn account, you will be paid \$15 for the baseline survey (plus being fully enrolled by joining the group), \$20 for completing the 4-week survey, and an additional \$15 if you show proof of at least the first dose of vaccination (send us picture of vaccine card). You will receive a total of \$50 if you complete all study questionnaires and tasks.
- There is no cost to you for participation in this study. However, there may be out-of-pocket expenses such as internet fees.
- All research data collected will be stored securely and confidentially (Names, dates, email addresses, phone numbers, facial images from Facebook/TikTok/ other social media profile photo, public photos/videos and IP addresses). Confidentiality will be maintained by means of having your responses coded so that they cannot be identified. The codes will be kept on a computer that will be stored securely. Only the investigator will have access to this information. Additionally, identifiers might be removed from the identifiable private information and, after such removal, the information could be used for future research studies without additional informed consent from you.
- The research team, authorized UCI personnel, and regulatory entities, may have access to your study records to protect your safety and welfare.

• While the research team will make every effort to keep your personal information confidential, it is possible that an unauthorized person might see it. We cannot guarantee total privacy.

#### Future Research Use

Researchers will use your information to conduct this study. Once the study is done using your information, we may share them with other researchers so they can use them for other studies in the future. We will not share your name or any other private identifiable information that would let the researchers know who you are. We will not ask you for additional permission to share this de-identified information.

• To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health (NIH). With this Certificate, researchers cannot be forced to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by NIH which is funding this project. You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law. Researchers will voluntarily disclose information to prevent serious harm to you or to someone else including, incidents of a child, elder, and dependent adult abuse or neglect, which will be reported to the appropriate authorities

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document. You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. It will be disclosed only with your permission. Identifiers collected (Names, dates, postal addresses, email addresses, phone numbers, facial images from Facebook profile photo, and IP addresses) will be removed before any potential future use for research studies without additional consent from you.

- The researchers intend to keep the de-identified research data indefinitely.
- ClinicalTrials.gov ClinicalTrials.gov is a Web site that provides information about clinical trials. A
  description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov/">http://www.clinicaltrials.gov/</a>, as required by U.S.
  Law. This Web site will not include information that can identify you. At most, the Web site will
  include a summary of the results. You can search this Web site at any time.
- Information collected from you for this study and/or information obtained from social networks (Facebook, TikTok, etc.) may be used in this research or other research, and shared with other organizations (de-identified data). You will not share in any commercial value or profit derived from the use of your information and/or information obtained from your social networks.

- If, during the course of this study, significant new information becomes available that may relate to your willingness to continue to participate, this information will be provided to you by the research team listed at the top of the form.
- If you have any comments, concerns, or questions regarding the conduct of this research please contact the researchers listed at the top of this form.
- It is important that you promptly tell the researchers if you believe that you have been injured because of taking part in this study. You can tell the researcher in person or call him/her at the number listed at the top of this form.
- Please contact the UCI Institutional Review Board by phone, (949) 824-7295, by e-mail at IRB@research.uci.edu or at 141 Innovation Drive, Suite 250, Irvine, CA 92697 if you are unable to reach the researchers listed at the top of the form and have general questions; have concerns or complaints about the research; have questions about your rights as a research subject; or have general comments or suggestions.
- If you have questions about your informed consent or any aspects of this consent form you can email your questions to hopecovid@hs.uci.edu.
- What is an IRB? An Institutional Review Board (IRB) is a committee made up of scientists and non-scientists. The IRB's role is to protect the rights and welfare of human subjects involved in research.
  The IRB also assures that the research complies with applicable regulations, laws, and institutional policies.

### **CONSENT OF STUDY PARTICIPANT**

I understand the procedures described above. My questions have been answered to my satisfaction.

Please print a copy of this page for your records

By clicking "Next", I agree to participate in the study.